CLINICAL TRIAL: NCT05136352
Title: Postoperative Analgesic Benefit of iPACK Block in the Anterior Cruciate Ligament Reconstruction Surgery, the LIGA-PACK Study
Brief Title: Postoperative Analgesic Benefit of iPACK Block in the Anterior Cruciate Ligament Reconstruction Surgery
Acronym: Liga-PACK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/21/0167; 2021-A01226-35 (Other: ID-RCB)
Record Dates: First submitted 2021-10-20; First posted 2021-11-29 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Anterior Cruciate Ligament Reconstruction
Keywords: loco-regional anesthesia; anterior cruciate ligament reconstruction; multimodal analgesia; motor sparing; iPACK block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adductor canal block (Active Comparator): loco-regional analgesia with adductor canal block (ACB) method (for anterior cruciate ligament reconstruction )
  Interventions: Procedure: adductor canal block
- iPACK block (Experimental): loco-regional analgesia with iPACK block (infiltration between the popliteal artery and the capsule of the posterior knee) ((for anterior cruciate ligament reconstruction )
  Interventions: Procedure: iPACK block

INTERVENTIONS:
Procedure: adductor canal block — loco-regional anesthesia using adductor canal block
  Other Names: ACB
  Arms: adductor canal block
Procedure: iPACK block — loco-regional anesthesia using infiltration between the popliteal artery and the capsule of the posterior knee
  Arms: iPACK block

SUMMARY:
This randomised clinical trial evaluates the analgesia provided by an iPack block associated with an adductor canal block in patients who undergo anterior cruciate ligament reconstruction surgery, compared to an adductor canal block alone. The objective is to prove the superiority of this locoregional anesthesia in terms of analgesia and functional rehabilitation.

DETAILED DESCRIPTION:
The ideal loco-regional anesthesia for anterior cruciate ligament reconstruction ensuring a satisfying analgesia without compromising an early rehabilitation is still undetermined.

Femoral nerve block has been incriminated in a delayed postoperative mobilization whereas the adductor canal block gives an equivalent analgesia for a better preservation of the quadricipital muscular strength.

The iPACK block (infiltration between the popliteal artery and the capsule of the posterior knee) is a recently described technique. Few studies have assessed the iPACK block in ACL reconstruction, and none were randomized.

This randomized single blind clinical trial compares two groups of 45 patients who undergo ACL reconstruction surgery under general anaesthetic : one receives an iPACK block associated with an adductor canal block, and the other only has an adductor canal block.

Pain scores and opioid consumption are collected after surgery in the recovery room, then by telephone interview at 24 and 48 hours post-surgery. Functional rehabilitation is evaluated by scales (KOOS, LYSHOLM and iKDC) at 3, 6 and 9 months after surgery. Adverse effects, due to anesthesia or opioids, are collected from 30 min after loco-regional anesthesia until the second phone call at 48h post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ACL repair surgery under general anesthesia
* Person affiliated or beneficiary of a social security plan
* Free, informed and written consent

Exclusion Criteria:

* Age < 18 years
* Contraindication to ALR (allergy to local anesthetics, local infection of the puncture site, coagulopathy)
* Pre-existing opiate dependence
* Contraindication to non-steroidal anti-inflammatory drugs
* Pregnant or potentially pregnant women
* Patients under the protection of adults (guardianship, curatorship or safeguard of justice)
* Patients whose cognitive state does not allow evaluation by the scales used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption at 48 hours after surgery | Hours 48
  Cumulative opioid consumption in the first 48 hours after anterior cruciate ligament repair surgery

SECONDARY OUTCOMES:
Cumulative opioid consumption at 2 hours after surgery | Hours 2
  Cumulative opioid consumption in the recovery room after anterior cruciate ligament repair surgery
Cumulative opioid consumption at 24 hours after surgery | Hours 24
  Cumulative opioid consumption in the first 24 hours after anterior cruciate ligament repair surgery
Cumulative opioid consumption at 3 months | month 3
  total opioid consumption at 3 months after anterior cruciate ligament repair surgery
Maximum pain score in the recovery room | hours 2
  Maximum pain score evaluated by the numerical pain scale from 0 to 10 (0 lowest pain score / 10 highest pain score)
Maximum pain score at 24 hours after surgery | hours 24
  Maximum pain score evaluated by the numerical pain scale from 0 to 10 (0 lowest pain score / 10 highest pain score)
Maximum pain score at 48 hours after surgery | hours 48
  Maximum pain score evaluated by the numerical pain scale from 0 to 10 (0 lowest pain score / 10 highest pain score)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice FERRE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

REFERENCES:
- [Derived] Ferre F, Boussaguet L, Vari N, Pillard F, Bosch L, Ferrier A, Ba C, Tissot B, Menut R, Kurrek M, Labaste F, Cavaignac E, Minville V. Comparison of femoral triangle plus iPACK blocks with femoral triangle block alone for anterior cruciate ligament reconstruction: a randomized controlled clinical trial on postoperative pain and knee function. Reg Anesth Pain Med. 2025 Mar 7:rapm-2024-106108. doi: 10.1136/rapm-2024-106108. Online ahead of print. PMID 40055004